CLINICAL TRIAL: NCT00849459
Title: Phase I Trial of Adenoviral Vector Delivery of the Human Interleukin-12 cDNA by Intratumoral Injection in Patents With Metastatic Breast Cancer
Brief Title: Gene Therapy in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Max Sung (Other)
Responsible Party: Sponsor-Investigator, Max Sung, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 02-0797; MTS-GCO-02-0797; NIH-0707-869; CDR0000629819
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adenovirus-mediated human interleukin-12 (Experimental): starting dose of ADV-hIL12 - 1 x 10 to the 10th power vp (virus particles) per patient, escalating in half-log increments up to 1 x 10 to the 13th power vp per patient, after which dose escalation will be at lower increments of 2 x 10 to the 13th power vp, to a maximum of 3.0 x 10 to the 13th power vp per patient.
  Interventions: Biological: adenovirus-mediated human interleukin-12

INTERVENTIONS:
Biological: adenovirus-mediated human interleukin-12 — The purified ADV-hIL12 is suspended in formulation buffer (10mM Tris, pH 7.5/
  1mM MgCl2/ 150mM NaCl/ 10% glycerol) and aliquoted into 1ml cryovials. The filled vials are stored at or below -60 degC.

SUMMARY:
RATIONALE: Placing the gene for interleukin-12 into breast cancer cells may help the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gene therapy in treating women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and maximum tolerated dose of intratumoral injection of adenovirus-mediated human interleukin-12 gene in women with metastatic breast cancer.
* Determine the tumor response in patients treated with this regimen.
* Determine the immune response in patients treated with this regimen.

OUTLINE: Patients receive a single dose of adenovirus-mediated human interleukin-12 intratumorally via percutaneous needle placement under ultrasound guidance.

Blood and tumor tissue samples are collected periodically for immunological laboratory studies. Samples are analyzed for serum cytokine levels by ELISA; qualitative analysis of immune biomarkers by IHC staining; and immune cell biomarker analysis by FACS.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the breast

  * Malignant disease in the skin, chest wall, or other sites (lymph nodes or primary tumor in the breast) accessible to percutaneous needle placement and injection

    * Solitary or multiple tumors
    * Measurable disease in ≥ 2 dimensions by physical examination or CT/MRI scan
    * Malignant tumors in the skin and chest wall must be ≥ 4 mm in diameter by physical examination
    * Malignant tumors in other accessible sites must be ≥ 1 cm in diameter on physical examination
  * Malignant disease in other organs (in addition to skin or chest wall metastases) allowed
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Karnofsky performance status 70-100%
* Life expectancy ≥ 16 weeks
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 mg/dL
* PT normal
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 45 mL/min
* Serum total bilirubin ≤ 2.0 times upper limit of normal (ULN)
* Serum transaminases ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Weight ≥ 30 kg (for patients treated with the highest dose level of study drug)
* No active infection or concurrent serious medical illness
* No HIV positivity
* No other malignancy within the past 5 years except for the following:

  * Inactive nonmelanoma skin cancer
  * In situ carcinoma of the cervix
  * Grade 1 papillary bladder cancer

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No anticoagulant therapy with heparin or warfarin for ≥ 2 months after completion of study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | up to 1 month
  Serum antibodies (titer) to adenovirus
Toxicity and safety | up to 2 months
  adverse events as assessed by NCI CTCAE v3.0

SECONDARY OUTCOMES:
Tumor response progression) | up to 2 months
  Sequential assessment of tumor on CT or MRI (complete response, partial response, stable disease, or disease)
Immune response | up to 2 months
  Serum IL12, and IFNγ levels. Serum antibodies (titer) to adenovirus.

CONTACTS AND LOCATIONS:
Overall Officials: Max W. Sung, MD, Principal Investigator — Icahn Medical Center at Mount Sinai
Locations (1):
- Icahn Medical Center at Mount Sinai, New York, New York, United States